CLINICAL TRIAL: NCT00388414
Title: Functional MRI Neural Correlates of Medication Efficacy in Patients With Chronic Low Back Pain
Brief Title: Imaging Study of Chronic Low Back Pain in Patients Taking Pain Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Redlich Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: F1J-MC-I006
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo - sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo
- Duloxetine (Experimental)
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — 30-60mg of duloxetine daily
  Arms: Duloxetine
Drug: Placebo — Placebo pill once daily
  Arms: Placebo - sugar pill

SUMMARY:
Duloxetine has recently been shown to be effective in reducing the pain in chronic pain patients. Duloxetine is known to exert a central mechanism, however the precise human brain structures responsible for mediating its pain-relieving properties are not known. We will use functional magnetic resonance imaging (FMRI) to investigate the neural and functional correlates of pain.

ELIGIBILITY:
Inclusion Criteria:- Males aged 18-60

* Back Pain
* Must be able to comply with study visit schedule and other study requirements
* Capable of performing the experimental tasks Exclusion Criteria:- Contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body)
* Known hypersensitivity to duloxetine or any of the inactive ingredients
* Uncontrolled narrow-angle glaucoma

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- See also: Description of the study and recruitment details — http://snapl.stanford.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Duloxetine: In the first 8-week treatment period, participants received placebo to match duloxetine for 8 weeks. Following a -week washout period, in the second 8-week treatment period, participants received duloxetine starting at 30 mg (1 week), with titer up to 60 mg (2 weeks), maintained dose (4 weeks), and titer back down to 30 mg (1 week).
- Duloxetine Then Placebo: In the first 8-week treatment period, participants received duloxetine starting at 30 mg (1 week), with titer up to 60 mg (2 weeks), maintained dose (4 weeks), and titer back down to 30 mg (1 week). Following a -week washout period, in the second 8-week treatment period, participants received placebo to match duloxetine for 8 weeks.
Period: First Intervention (8 Weeks)
Arm/Group | Placebo Then Duloxetine | Duloxetine Then Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo Then Duloxetine | Duloxetine Then Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Placebo Then Duloxetine | Duloxetine Then Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Duloxetine | Duloxetine Then Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11.36) | 42.86 (12.56) | 36.93 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Brief Pain Inventory (BPI) scores were obtained at baseline, weeks 1, 2, 6, 7, 8, and 12, and a follow-up visit one week after completing the study.
  Responses are rated on a scale from 0-10, with 0 = no pain and 10 = pain as bad as you can imagine.
  Placebo and duloxetine pain scores calculated by averaging pain scores from each visit after baseline.
  Values were converted to percent change in pain: [(baseline pain - end point pain)/baseline pain] x 100.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Percentage change from baseline to end
Arm/Group | Placebo - Sugar Pill | Duloxetine
Number analyzed (Participants) | 14 | 14
Percentage change from baseline to end | -1 (76) | -43 (32)

2. Primary Outcome: Neural Correlates of Pain Relief
Description: Scores reflect the average connectivity strength of that region of interest to the rest of the cortex.
  There were no minimum or maximum values on this scale. Higher scores reflect stronger connectivity, and lower scores reflect less connectivity (all scores fell within -3 and 3).
  Subscales are averaged.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Baseline: Pre-treatment
Arm/Group | Baseline | Placebo - Sugar Pill | Duloxetine
Number analyzed (Participants) | 14 | 14 | 14
Units on a scale
  Ventral Default Mode Networks | 0.521 (0.346) | 0.466 (0.279) | 0.468 (0.443)
  Dorsal Default Mode Networks | 0.485 (0.277) | 0.492 (0.203) | 0.469 (0.315)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of the study, for 12 weeks.
Description: The clinicaltrials.gov definition of adverse event and/or serious adverse event was used to collect adverse event information.
Groups:
- All Participants: Includes all participants.
  Placebo: Placebo pill once daily Duloxetine: 30-60mg of duloxetine daily
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No